CLINICAL TRIAL: NCT06432634
Title: Effects of Comprehensive Pulmonary Rehabilitation Programs (CPRP) on Patients Undergoing Lung Resection: a Randomized Controlled Trial
Brief Title: Effects of CPRP on Patients Undergoing Lung Resection
Acronym: CPRP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202400512B0
Record Dates: First submitted 2024-05-12; First posted 2024-05-29 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-05

CONDITIONS: Rehabilitation
Keywords: lung resection surgery; comprehensive pulmonary rehabilitation programs; six-minute walk test; quality of life; biomarkers
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Masking Description: The blinding of patients to their treatment group allocation is unattainable owing to the inherent nature of the exercise intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard care group (Sham Comparator): Participants randomize to the standard care group (SC) receive the standard care already established in Chiayi Chang Gung Memorial Hospital. Standard care comprises one therapeutic education session conducted by a respiratory therapist 1-2 weeks before surgery.
  Interventions: Other: Standard care
- comprehensive pulmonary rehabilitation program group (Experimental): Participants randomize to the comprehensive pulmonary rehabilitation program group (CPRP) undergo an evidence-based and hospital-based comprehensive pulmonary rehabilitation program developed by the research group. This program is administered in addition to the standard care provided and spans across the preoperative, peri-operative, and postoperative periods, covering a total of 1-2 weeks preoperatively and 3-6 weeks postoperatively. CPRP involves warm-up and cool-down exercises, the aerobic training, and the resistance training. Additionally, participants are encouraged to continue exercising at home or in community sports facilities.
  Interventions: Other: Standard care; Other: Comprehensive pulmonary rehabilitation programs

INTERVENTIONS:
Other: Standard care — The pre-operative educational session has a duration of 40 minutes and covers pre-operative education, breathing exercises (diaphragmatic breathing, deep breathing techniques and sustained maximal inflation), and airway clearance techniques (directed cough, huffing, and chest physiotherapy). Patients are instructed to perform these techniques ten times per waking hour, every day. The in-patient peri-operative session incorporates intermittent positive pressure breathing inhalation (IPPB) administered for 15 minutes twice daily. Inhalation therapy involving mucolytics and bronchodilators is administered three times per day, and early mobilization is encouraged until discharge. Upon discharge, participants are encouraged to continue practicing breathing exercises, deep breathing techniques, and maintaining an active level of activity.
Other: Comprehensive pulmonary rehabilitation programs — 1. Warm-up and cool-down exercises: stretching various muscle groups for a duration of 15 to 20 minutes and a slow 3-minute walk
  2. Aerobic training: using a lower-limb cycle ergometer for a duration of 30 to 40 minutes. Initiated warm-up at 0 wattages for 5 minutes. Incrementally increased wattages within 5-10 minutes until reaching the 40-80% heart rate reserve or 4 to 6 of modified Borg scale for at least 20 minutes. Concludes with a 5-minute cool-down period at 10 wattages.
  3. The resistance training involves both upper and lower limbs:
  （1） Upper Limb Resistance Training: Shoulder lift, abduction, and horizontal abduction exercises are performed. Each exercise is repeated for three sessions comprising 10 repetitions each. A 0.5-2 kg dumbbell is utilized for resistance.
  （2） Lower Limb Resistance Training: Sit-to-stand exercises are performed. Each session consists of three sets of 10 repetitions.
  Arms: comprehensive pulmonary rehabilitation program group

SUMMARY:
The aim of this project is to investigate the effectiveness of implementing a Comprehensive Pulmonary Rehabilitation Program (CPRP) in patients undergoing lung resection surgery. The CPRP encompasses a training regimen combining aerobic exercise, resistance exercises, breathing exercises, and home activities, specifically tailored for patients with limited exercise capacity and impaired lung function. The study seeks to understand the physiological and biological effects of the CPRP in this patient population.

DETAILED DESCRIPTION:
Background: Elderly patients with compromised lung function or poor health conditions undergoing lung resection surgery face an increased risk of postoperative pulmonary complications. Pulmonary rehabilitation programs play a crucial role in enhancing recovery after surgery, having been shown to reduce postoperative pulmonary complications and enhance patients' pre- and post-operative exercise capacity, functional performance, and quality of life. However, due to the heterogeneity of interventions in pulmonary rehabilitation programs, the optimal timing, methods, or duration of exercise training for lung resection patients remain unclear. Additionally, there is a lack of comprehensive research on the changes and impacts of biomarkers in the blood of lung resection patients following intervention with pulmonary rehabilitation programs.

Objectives: This study aims to investigate the physiological and biological effects of a comprehensive pulmonary rehabilitation program in lung resection surgery patients with limited exercise capacity and impaired lung function.

Research Methods: This study adopts an open label, randomized, parallel design, intending to recruit 96 lung resection surgery participants divided into a control group receiving standard care and an experimental group receiving the comprehensive pulmonary rehabilitation programs. The intervention period spans 1-2 weeks pre-surgery, during hospitalization, and 3-6 weeks post-discharge. Participants will undergo four assessments at randomization (baseline, T0), one day pre-surgery (T1), the day of discharge post-surgery (T2), and at trial completion (T3). The primary endpoint is the six-minute walk test. Secondary endpoints include lung function, lung expansion volume, respiratory muscle strength, incidence of postoperative complications and pulmonary complications, chest tube duration, length of hospital stay, quality of life (EORTC QLQ-C30), and pain. Exploratory endpoints involve inflammation-related and immune-related biomarkers.

Expected Impact: This study will provide valuable insights into the physiological and biological effects of a comprehensive pulmonary rehabilitation programs for lung resection surgery patients. Results may contribute to improving patient outcomes and advancing academic understanding and clinical guidelines in this field.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥ 20 years old)
* Receiving lung resection surgery
* At least one of the following:

  6MWD < 500 meters, oxygen saturation by pulse oximetry (SpO2) drop ≥ 4% or SpO2< 90% during 6MWT, pre-operative forced expiratory volume in 1 second (FEV1) or forced vital capacity (FVC) ≤ 80% of predicted value or FEV1/FVC ratio ≤ 0.7
* Able to walk autonomously without mobility aids
* Written informed consent

Exclusion Criteria:

* Neoadjuvant therapy with chemo- or radiotherapy in the six months prior to surgery
* Received pulmonary rehabilitation programs six months prior to surgery
* Previous lung resection
* Inability to perform the exercise training
* Instability in cardiovascular disease, neurological disorders, or musculoskeletal conditions
* Have cognitive deficits with potential severe impact on compliance
* Do not provide written informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Six-minute walk distance (6MWD) | Baseline; one day pre-surgery; an average of post-surgery 2 weeks; through study completion, an average of 10 weeks
  Six-minute walk test (6MWT) is a sub-maximal exercise test used to assess aerobic capacity and endurance.

SECONDARY OUTCOMES:
Pulmonary function test | Baseline; one day pre-surgery; an average of post-surgery 2 weeks; through study completion, an average of 10 weeks
  Using spirometry to measure pulmonary function parameters.
Respiratory muscle strength | Baseline; one day pre-surgery; an average of post-surgery 2 weeks; through study completion, an average of 10 weeks
  Measurement of respiratory muscle strength includes maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP), which assess the force exerted by muscles during maximal inspiratory and expiratory efforts, respectively. During the test, the subject sits and uses a mouthpiece connected to an electronic pressure gauge while wearing a nose clip to prevent air leakage. For MIP, the subject starts from residual volume and performs a maximal inspiratory effort. For MEP, the subject starts from total lung capacity and performs a maximal expiratory effort. The highest value from three measurements is recorded as the test result.
Length of hospital stay (LoS) | an average of post-surgery 2 weeks
  Length of hospital stay
Duration of chest-tube insertion | an average of post-surgery 2 weeks
  Duration of chest-tube insertion
Numerical Rating Scale (NRS) | Baseline; one day pre-surgery; an average of post-surgery 2 weeks; through study completion, an average of 10 weeks
  The Numerical Rating Scale (NRS) is a commonly used clinical tool for assessing pain intensity, ranging from 0 to 10 to represent varying degrees of pain. It is scored from 0-10 (0 meaning no pain and 10 meaning the worst pain.
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30, version 3, Chinese Mandarin (Taiwan)) | Baseline; one day pre-surgery; an average of post-surgery 2 weeks; through study completion, an average of 10 weeks
  The EORTC QLQ-C30 is designed to assess health-related quality of life in cancer patients, consisting of 30 items. It includes five functional scales: cognitive (2 items), emotional (4 items), physical (5 items), role (2 items), and social (2 items) functions. Symptom scales cover fatigue (3 items), nausea/vomiting (2 items), and pain (2 items). Single items assess appetite loss, constipation, diarrhea, dyspnea, sleep disturbances, and financial difficulties. Additionally, two items evaluate overall health status/quality of life. Each item is equally weighted, with scores linearly transformed to a 0-100 scale. For functional scales and overall health status/quality of life, higher scores indicate better function or quality of life, whereas higher scores on symptom scales denote more severe symptoms or problems.
Postoperative complications (POCs) and postoperative pulmonary complications (PPCs) | an average of post-surgery 2 weeks
  Postoperative complications (POCs) and postoperative pulmonary complications (PPCs)
Lung expansion volume | Baseline; one day pre-surgery; an average of post-surgery 2 weeks; through study completion, an average of 10 weeks
  measured by volume-oriented incentive spirometry

OTHER OUTCOMES:
inflammation-related and immune-related biomarkers | Baseline; one day pre-surgery; an average of post-surgery 2 weeks; through study completion, an average of 10 weeks
  insulin-like growth factor-1 (IGF-1), insulin-like growth factor binding protein-3 (IGFBP-3), C reactive protein (CRP), Surfactant Protein-D (SP-D), Granulocyte-macrophage colony-stimulating factor (GM-CSF), interleukin (IL)-1 beta, IL-2, IL-4, IL-5, IL-6, IL-10, IL-12 p70, IL-13, IL-18, tumor necrosis factor (TNF)-alpha, interferon (IFN)-gamma

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Jung Chang, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: No